CLINICAL TRIAL: NCT01387945
Title: Pilot Study of Home Blood Pressure Control Program (eBP Control)
Acronym: eBPcontrol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Hospital of Rhode Island (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Charles B. Eaton, Director of Center for Primary Care and Prevention, Memorial Hospital of Rhode Island
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: NCT 01242319; 1R21HS018238-01 (AHRQ)
Record Dates: First submitted 2011-07-01; First posted 2011-07-06 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Hypertension; Cardiovascular Disease
Keywords: Home blood pressure monitoring; Patient activation; Patient-centered care; Community Health Aides; Primary Health Care
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Patient Participation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HBPM only (No Intervention)
- HBPM+website+patient navigator (Experimental)
  Interventions: Behavioral: HBPM+website+patient navigator

INTERVENTIONS:
Behavioral: HBPM+website+patient navigator — In addition to home blood pressure monitor, patient receives access to BP web portal and trained patient navigator.
  Other Names: Good Health Gateway
  Arms: HBPM+website+patient navigator

SUMMARY:
This intervention study will evaluate the feasibility,acceptability and effectiveness of an e-health enabled model of care by randomly assigning a trained patient navigator and/or a blood pressure (BP) self-management web portal to patients with uncontrolled hypertension after a run in period with a home BP monitor (HBPM) and comparing the results on blood pressure control. We anticipate that patients receiving the combination of a patient navigator(PN)with a self-management web portal and home BP monitor will have better BP control than when the only received a home BP monitor.

DETAILED DESCRIPTION:
The study will demonstrate and evaluate the feasibility and acceptability of an e-health enabled model of care for improved hypertension and elevated blood pressure control using a home blood pressure monitor (HBPM), a blood pressure (BP) self-management web portal, and a trained patient navigator. During the first or the control period, all of the participants will have access to the only the HBPM. The control period will be compared to the final or the intervention period when the participants will gain access to a trained patient navigator and the web portal. This comparison will assist in estimating the effect sizes of the HBPM plus PN plus self-management web portal to HBPM alone for each of the outcomes: patient activation, self-management activities, medication adherence, reduced clinical inertia, and improved BP control. The second of the randomization periods will allocate a patient navigator to half of the participants, while the other half will gain access to only the web portal. We will compare the effectiveness of the PN plus webportal plus HBPM to webportal plus HBPM during this second period. An evaluation of the intervention process will delineate the barriers and facilitators by the providers, participants, and patient navigators.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed w/ hypertension or elevated blood pressure, uncontrolled blood pressure at the baseline research visit according to the following risk levels:

  * Average risk,
  * SBP >140 mmHg or DBP > 90 mmHg;
* Vascular disease (cerebrovascular disease, coronary heart disease, diabetes mellitus, peripheral vascular disease, renal insufficiency)
* SBP >130 mmHg or DBP >80 mmHg;
* Left ventricular dysfunction,
* SBP 120 mmHg or DBP >80 mmHg;
* can read and understand English; must have access to internet

Exclusion Criteria:

* Unable to comply with protocol;
* pregnancy;
* secondary hypertension (e.g. renovascular);
* participation in other hypertension clinical trials;
* hospitalized in the past six months for diabetes, renal failure, or heart failure;
* severe renal insufficiency (estimated glomerular filtration rate < 30 mL/min);
* patient already routinely using a home blood pressure monitoring device or patient not able to use HBPM device due to disability;
* arm circumference larger than 17 inches determined during telephone screener,
* arm circumference smaller than 9 inches measured at baseline research visit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-09; Primary Completion 2012-05 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Percent of patients at BP goal | Nine months
  Percentage of patients at systolic and/or diastolic blood pressure at goal at the fourth research visit (end of the study)

SECONDARY OUTCOMES:
Health status | Nine Months
  SF-12 questionnaire, patient activation
Use of intervention tools | Nine months
  home blood pressure monitor-amount of time at goal; number of times patient utilized the website
Costs | Nine months

CONTACTS AND LOCATIONS:
Overall Officials: Charles B Eaton, MD, Principal Investigator — Memorial Hospital of Rhode Island
Locations (1):
- Memorial Hospital of Rhode Island, Pawtucket, Rhode Island, United States